CLINICAL TRIAL: NCT04304339
Title: Hypercapnic Acute Respiratory Failure in the ICU : the YETI Study
Acronym: YETI
Status: Completed | Type: Observational
Sponsor: French Society for Intensive Care (Other)
Responsible Party: Sponsor
Other Study IDs: YETI
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Intensive Care Unit Syndrome; Hypercapnia; Acute Respiratory Failure
MeSH Terms: conditions — Hypercapnia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Hypercapnic respiratory failure — Patients with hypercapnic respiratory failure will be followed without any additional intervention

SUMMARY:
Hypercapnia is a frequent clinical situation defined as an elevation of the partial pressure of carbon dioxide (PaCO2) above 45 mmHg. Several physiopathological parameters such as respiratory minute volume, dead space volume or CO2 production influence the PaCO2. Therefore, hypercapnia can affect the time of various diseases.

Available epidemiological data regarding hypercapnia are from studies investigating the efficacy of non-invasive ventilation (NIV), with different population cohorts. However, their interpretation must be cautious given the heterogeneity in patient case-mix and results.

Then, whether hypercapnia is a common reason for intensive care unit (ICU) admission, epidemiological data is scarce and heterogeneous. The aim of this study is to investigate the epidemiological, clinical determinants and outcomes of patients admitted to ICU with hypercapnic respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥18 years old presenting with at least of the following items :

  1. respiratory rate ≥ 25/min,
  2. paradoxical motion of the abdomen,
  3. intercostal retraction AND
* a PaCO2 > 45 cm H20 before ICU admission or within the 12 hours following ICU admission.

Exclusion Criteria:

* Refusal to give informed consent,
* pregnancy,
* < 18 years patient,
* dying patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The aim of this study is to investigate the epidemiological, clinical determinants and outcomes of patients admitted to ICU with hypercapnic respiratory failure.
Sampling Method: Probability Sample
Enrollment: 862 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Prevalence of hypercapnic acute respiratory failure in ICU | Intensive Care Unit length stay (Usually 7 days)
  Number of patients with hypercapnic acute respiratory failure in ICU related to number of patients admitted in the ICU during study period

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CH Andre Migniot, Versailles, A
  - CHU Nantes, Nantes
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided